CLINICAL TRIAL: NCT05548517
Title: Time Restricted Eating on the Microbiome Affecting Metabolic Health and Bone in Older Women
Brief Title: TRE: Microbiome, Metabolic Health and Bone
Acronym: TREMBO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sue A. Shapses, Ph.D., RD, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021002434
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Weight Loss; Time Restricted Feeding; Bone Loss
Keywords: bone mineral density; Microbiome; obesity and overweight; metabolic health; time restricted feeding; energy restriction
MeSH Terms: conditions — Weight Loss; Intermittent Fasting; Bone Diseases, Metabolic; Obesity; Overweight | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
  Enroll 48 to achieve sample size of 40 (20/group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted eating and calorie restriction (Experimental): Subjects will be asked to adhere to a calorie-restricted diet and will be counseled by a dietitian for diet and lifestyle behavior education. In addition, they will be asked to only consume calories during a 9-hour window (15:9).
  Interventions: Behavioral: Time Restricted Eating (TRE); Behavioral: Calorie Restriction
- Calorie restriction alone (Active Comparator): Subjects will be asked to adhere to a calorie-restricted diet and will be counseled by a dietitian for diet and lifestyle behavior education. They will be advised to continue to consume foods throughout the day and into the evening.
  Interventions: Behavioral: Calorie Restriction

INTERVENTIONS:
Behavioral: Time Restricted Eating (TRE) — 9-hour eating window
  Arms: Time restricted eating and calorie restriction
Behavioral: Calorie Restriction — daily calorie restriction

SUMMARY:
In the Time-Restricted Eating: Microbiome and Bone (TREMBO) study, the primary goal is to determine the effect of time-restricted eating with caloric restriction compared to caloric restriction alone on body weight, the gut microbiota, and bone health in older women who are overweight or obese.

DETAILED DESCRIPTION:
Time-restricted eating (TRE) has gained increased attention due to the possibility to induce weight loss and improve cardiometabolic health as a result of the purported alignment of circadian rhythm. However, since TRE is often reported to cause a spontaneous reduction of calories, it is not well understood if these health benefits are due to weight loss, circadian rhythm alignment, or a combination of the two. Furthermore, while weight loss can improve cardiometabolic health, it can also induce bone loss, which is problematic in older women who are at a higher risk of fracture. Interestingly, both bone turnover and the gut microbiota are responsive to diurnal variations, such as meal timing, and alterations in the gut microbiota have been associated with differences in bone health. In rodent models, caloric restriction can alter the gut microbiota composition with further alterations shown due to time-restricted eating. This suggests that time-restricted eating could affect bone health, which may be partially mediated by changes in the gut microbiota. Also, lifestyle patterns affects both the microbiota and bone. This randomized controlled trial will use behavior modification to examine TRE plus caloric restriction (CR) to achieve an evening energy deficit compared to CR alone on body weight, the gut microbiota, and bone health in older women who are overweight or obese.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (>2 years since last menses)
* Body mass index (25-45 kg/m2)
* Agree to be randomly assigned to consume food for ≤ 9 hours/day or ≥12 hours/day
* Must attend on-site visits (about 10) in New Brunswick, NJ, USA (transportation/reimbursement for travel not included)

Exclusion Criteria:

* Participants with >5% weight loss in the past 6 months or extreme dietary/physical activity habits
* An inability to follow the experimental intervention or to perform the required specimen collections
* Antibiotic use in the past 2 months
* Current diagnosis, or history of cancer in past 3 years
* History of surgical procedure for weight loss in the past 3 years
* Current diagnosis or history of bone diseases, type I or II diabetes, gastrointestinal disease, hyperparathyroidism, untreated thyroid disease, significant immune, hepatic, cardiac, or renal disease
* Uncontrolled hypertension or hyperlipidemia in abnormal ranges
* Regular use of medications that affect bone metabolism, including bisphosphonates or hormone replacement.
* A colonoscopy within the past 2 months
* Alcohol or illicit drug abuse
* Current smoker or having quit smoking in the past 3 months
* Shift work
* Participation in another clinical research trial which may interfere with the results of this study.

Ages: 50 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 48 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss | change from baseline to an average 6 months
  Body weight in kg
Bone mineral density (BMD - hip) | change from baseline to an average 6 months
  dual energy x-ray absorptiometry
Microbiota | change from baseline to an average 6 months
  stool

SECONDARY OUTCOMES:
Soft tissue (lean and fat mass) | change from baseline to an average 6 months
  dual energy x-ray absorptiometry
Areal BMD (lumbar spine, femoral neck, radius, total body) | change from baseline to an average 6 months
  dual energy x-ray absorptiometry
Trabecular bone (volumetric BMD, bone volume / total volume, and separation) | change from baseline to an average 6 months
  peripheral quantitative computed tomography
Cortical bone (volumetric BMD, thickness, and porosity) and total BMD | change from baseline to an average 6 months
  peripheral quantitative computed tomography
Blood pressure (systolic and diastolic) | change from baseline to an average 6 months
  sphygmomanometer
Glucose - response to oral glucose tolerance test | change from baseline to an average 6 months
  fasting and response to glucose solution
Insulin - response to oral glucose tolerance test | change from baseline to an average 6 months
  fasting and response to glucose solution

OTHER OUTCOMES:
25-hydroxyvitamin D (25OHD) | change from baseline to an average 6 months
  serum
estradiol | change from baseline to an average 6 months
  serum
parathyroid hormone (PTH) | change from baseline to an average 6 months
  serum
Fasting osteocalcin | change from baseline to an average 6 months
  serum bone formation and energy marker
Fasting procollagen type 1 N-terminal propeptide (PINP) | change from baseline to an average 6 months
  serum bone formation marker
Fasting C-telopeptide of type I collagen (CTX) | change from baseline to an average 6 months
  serum bone resorption marker
Cognitive function | change from baseline to an average 6 months
  Cambridge Neuropsychological Test Automated Battery
melatonin | change from baseline to an average 6 months
  serum
cortisol | change from baseline to an average 6 months
  serum
Quality of sleep | change from baseline to an average 6 months
  Pittsburgh sleep quality index (0-21; higher score is worse)
Diet quality score | change from baseline to an average 6 months
  nutrient analysis software (Healthy Eating Index 0-100; higher score is better)
Eating self-efficacy | change from baseline to an average 6 months
  Weight lifestyle efficacy questionnaire short-form (0-80; higher score is better)
Circumferences | change from baseline to an average 6 months
  tape measure (waist, hip and thigh)
Short physical performance battery (SPPB) | change from baseline to an average 6 months
  Total score of SPPB (0-12; higher score is better)
6 minute walk test | change from baseline to an average 6 months
  total distance
Timed up and go | change from baseline to an average 6 months
  total time
Hand Grip | change from baseline to an average 6 months
  dynanometer (isometric grip force)

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University - NJ Inst Food Nutrition & Health, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No